CLINICAL TRIAL: NCT05999695
Title: Effects of the Self-management on Anxiety, Depression, Quality of Life and Self-management of Patients With Acute Coronary Syndromes: a Randomized Controlled Trial.
Brief Title: Self-management of Patients With Acute Coronary Syndromes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Cheng, Hui- Chuan, Nursing Supervisor, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022-08-003C
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Acute Coronary Syndromes
Keywords: self-management; acute coronary syndrome; anxiety; depression; quality of life
MeSH Terms: conditions — Acute Coronary Syndrome; Anxiety Disorders; Depression | interventions — Self-Management

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- self-management interventions (Experimental): self-management interventions: According to the results of literature search and based on the theory of self-efficacy, the intervention measures of the self-management program were designed.
  regular care:regular care
  Interventions: Other: self-management; Other: regular care
- regular care (Active Comparator): regular care
  Interventions: Other: regular care

INTERVENTIONS:
Other: self-management — The experimental group received the "SelfManagement Program for Acute Coronary Syndrome":
  the research subjects completed the first data collection within one week of hospitalization. Guide the research subjects to browse this manual and watch the "Acute Coronary Self-Care Video", and explain what they do not understand, hoping to stimulate the research subjects to discuss nursing issues, and jointly formulate self-management goals, and This handbook was given to study subjects to take home. Telephone interviews every 2 weeks in the first month after discharge, and then again after two and three months after discharge. Each call is about 10 minutes to track the completion of goals and self-management,including usual medication, regular exercise, balance Food and spiritual support and encouragement, etc.,and clarify any doubts.
  Arms: self-management interventions
Other: regular care — gular care regular care The nurse implements routine nursing instructions, including disease and treatment profiles,symptom management, and outpatient follow-up. Scan the QRC with your mobile phone or provide the "Care Guidance Leaflet for Coronary Artery Disease" and "Caring for Myocardial Infarction Patients" which are all written in text.

SUMMARY:
Purpose :

The purpose of this study is to investigate the tracking effect of selfmanagement programs on anxiety, depression, and quality of life in patients with Acute Coronary Syndromes (ACS).

DETAILED DESCRIPTION:
Research Design :

This study the first phase is to construct and develop interventional measures for self-management of patients with ACS. According to the associated factors of study, the intervention measures are designed based on self-management. A pilot study will be conducted to improve research and to develop better selfmanagement interventions in the future. At the secondary stage: a randomized controlled trial with a random sampling design is used to investigate the effects of self-management programs on anxiety, depression, and quality of life in patients with ACS. The study will conduct in a cardiac medicine ward or coronary intensive care center of a north medical center. Patients with ACS,who met the conditions and agreed to join the study will be recruited. Then,the informed consent will be obtained. At the first stage, 10subjects will be collect. At the secondary stage, a total of 104 subjects will be enrolled, 52 in the experimental group will receive the self-management program, and 52 in the control group will receive a routine hospital care.

Method & Results:

The data of demographic and disease characteristics, clinical indicators,depression, anxiety, self-management, and quality of life will be collected.The Hospital Anxiety and Depression Scale, the SF-36 Taiwan version of the Quality-of-Life Questionnaire and the Self-Management Scale will used as tools to collect data. The efficacy of the intervention will be collected 1 month and 3 months after the intervention. Data will be statistically analyzed by GEE.

Hypothesis :

It is expected that the self-management program applied to patients with ACS can reduce depression and anxiety, thereby improving the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Over 20 years old
* The first diagnosis of acute coronary syndrome by a clinician,
* Clear consciousness, able to converse in Chinese and Taiwanese languages.
* Willingness to participate in this research

Exclusion Criteria:

* Those who are unable to take care of themselves
* Poor vision and inability to read
* Hard of hearing and deafness
* Inability to communicate

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-12-11 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08-26 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale, HADS | First time(baseline) is in the first day in the ward.The second time is one month after discharge.The third time is three months after discharge.
  The Likert four-point scale (0-3 points) was used, and the two items were scored separately, and the total score was between 0-21 points. The higher the score, the higher the degree of anxiety or depression. A score below 7 means no anxiety or depression, a score between 8 and 10 means the patient is suspected of anxiety or depression, and a score greater than or equal to 11 means that the patient has anxiety or depression.
  It is a measure to assess change at three-time points. change from Baseline Anxiety and Depression at 1 and 3 months.
The MOS 36-Item Short-Form Health Survey,SF36 | First time(baseline) is in the first day in the ward.The second time is one month after discharge.The third time is three months after discharge
  Scores range from 0 to 100, with higher scores indicating better self-assessed health. Each item of the questionnaire is calculated separately according to the designed initial scores. Then the scores of the items related to each scale are added up and then subtracted from each scale to obtain the lowest score. Divide by the distance between the possible scores of each scale, and multiply by 100 to get the score.
  It is a measure to assess change at three-time points. change from Baseline quality of life at 1 and 3 months.
The Partner In Health scale, PIH | First time(baseline) is in the first day in the ward.The second time is one month after discharge.The third time is three months after discharge
  Items in the scale are graded on a nine-point scale, with 0 representing the worst and 8 representing the best. This is a closed and continuous variable. The scale scores range from 0 to 96, with higher scores indicating better selfmanagement.
  It is a measure to assess change at three-time points. Change from self-management Baseline at 1 and 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chuan Cheng, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei County,, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bandura, A. (1977). Self-efficacy: toward a unifying theory of behavioral change. Psychological Review, 84(2), 191-215. https:// doi.org/10.1037//0033-295x.84.2.191 Gach, O., El, H. Z., & Lancellotti, P.(2018). [Acute coronary syndrome]. Revue Médicale de Liège, 73(5-6),243-250. (Syndrome coronarien aigu.) Guo, P., & Harris, R. (2016). The effectiveness and experience of self-management following acute coronary syndrome: A review of the literature. International Journal of Nursing Studies,61, 29-51. https://doi.org/10.1016/j.ijnurstu.2016.05.008 Hong, P. C., Chen,K. J., Chang, Y. C., Cheng, S. M., & Chiang, H. H. (2021). Effectiveness of Theory-Based Health Information Technology Interventions on Coronary Artery Disease Self-Management Behavior: A Clinical Randomized Waitlist-Controlled Trial. Journal of Nursing Scholarship, 53(4), 418-427. https://doi.org/10.1111/ jnu.12661